CLINICAL TRIAL: NCT00827086
Title: Evaluation of Influencing Factors in Uveitis
Brief Title: Influencing Factors in Uveitis
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Eyeclinic, St Franziskus Hospital
Other Study IDs: 2008-089-f-S
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Uveitis
Keywords: influencing factors (smoking, nutrition, education)
MeSH Terms: conditions — Uveitis; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with non-infectious Uveitis
- 2: Patients with scleritis

SUMMARY:
Environmental factors possibly influencing uveitis are evaluated.

DETAILED DESCRIPTION:
Smoking, nutrition, BMI, education

ELIGIBILITY:
Inclusion Criteria:

* Patients with Uveitis

Exclusion Criteria:

* Children under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Uveitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-03; Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Heiligenhaus, Prof, MD, Study Chair — Department of Ophthalmology at St. Franziskus Hospital; Martin Rösel, MD, Principal Investigator — Department of Ophthalmology at St Franziskus Hospital Muenster
Locations (1):
- Department of Ophthalmology at St. Franziskus Hospital, Münster, Northrhine-Westfalia, Germany

REFERENCES:
- [Derived] Roesel M, Ruttig A, Schumacher C, Heinz C, Heiligenhaus A. Smoking complicates the course of non-infectious uveitis. Graefes Arch Clin Exp Ophthalmol. 2011 Jun;249(6):903-7. doi: 10.1007/s00417-010-1597-1. Epub 2011 Jan 5. PMID 21207052